CLINICAL TRIAL: NCT04441177
Title: Effects of PlayStation®VR on the Health-Related Quality of Life in Stroke Patients Undergoing Inpatient Rehabilitation: a Pilot Study
Brief Title: Effects of PlayStation®VR on the HRQOL in Stroke Patients Undergoing Inpatient Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Min Chen, Principal Investigator, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201801607A3
Record Dates: First submitted 2020-06-16; First posted 2020-06-22 (Actual); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Stroke
Keywords: Stroke; Virtual Reality; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: All participants are randomly allocated to study group and control group. Each participant's main study period is set as 16 days with additional follow-up time at post-intervention 3 months. Participants in the control group receive conventional rehabilitation therapy over 50 minutes on weekdays. Participants in the study group receive conventional rehabilitation therapy over 50 minutes on weekdays and 7 sessions (flexible schedule in different day) of PlayStation®VR of 20 minutes each in the main 16-day study period.
Who Masked: Outcomes Assessor
Masking Description: Pre-intervention, post-intervention, and 3-month follow-up HRQOL will be assessed by the Stroke Impact Scale (SIS) 3.0. Motricity Index (MI) and Fugl-Meyer Assessment (FMA), Functional Independence Measure (FIM), and arm movement ratio (AMR) will also be checked before intervention, after intervention, and at 3-month follow-up. One blinded occupational therapist will evaluate the outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Participants in the study group receive conventional rehabilitation therapy over 50 minutes on weekdays and 7 sessions (flexible schedule in different day) of PlayStation®VR of 20 minutes each in the main 16-day study period.
  Interventions: Device: PlayStation®VR training
- Control group (No Intervention): Participants in the control group receive conventional rehabilitation therapy over 50 minutes on weekdays.

INTERVENTIONS:
Device: PlayStation®VR training — Participants in the study group receive conventional rehabilitation therapy over 50 minutes on weekdays and 7 sessions (flexible schedule in different day) of PlayStation®VR of 20 minutes each in the main 16-day study period.
  Arms: Study group

SUMMARY:
Compared to conventional rehabilitation therapy, the full-immersive commercial game (CG) system, in the form of available video game, could safely provide more positive effect on health-related quality of life (HRQOL) and motor function in post-stroke patients.

The study aims to perform the research from 2019/7/1 to 2021/6/30 and enrolls a total of 80 participants. Stroke participants are recruited from the rehabilitation ward of CGMH hospital.

The inclusion criteria are (a) first-time unilateral cerebral stroke, (b) stroke onset less or equal to 1 year, (c) admission to the rehabilitation ward, (d) ages 20-80 years, (e) spasticity of paretic arm ≤ grade 2 in the Modified Ashworth Scale, and (f) no active medical problems such as fever, pneumonia, or scabies. The exclusion criteria are (a) brainstem or cerebellar stroke, (b) epilepsy history, including photosensitive epilepsy, (c) previous or active heart diseases, such as myocardial infarction or angina, (d) visuospatial problems related to stroke, such as hemianopia or hemineglect, (e) paretic upper limb reaches Brunnstrom recovery stage VI, (f) severe aphasia, (g) severe cognitive impairment, and (h) poor cooperation with assessments.

All participants are randomly allocated to study group and control group. Participants in the control group receive conventional rehabilitation therapy over 50 minutes on weekdays. Participants in the study group receive conventional rehabilitation therapy over 50 minutes on weekdays and 7 sessions (flexible schedule in different day) of PlayStation®VR of 20 minutes each in the main 16-day study period. Pre-intervention, post-intervention, and 3-month follow-up HRQOL will be assessed by the Stroke Impact Scale 3.0. Motricity Index and Fugl-Meyer Assessment, Functional Independence Measure, and arm movement ratio will also be checked before intervention, after intervention, and at 3-month follow-up. The safety outcome, intervention-related adverse events or any serious adverse events, during study period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* first-time unilateral cerebral stroke
* stroke onset less or equal to 1 year
* admission to the rehabilitation ward
* ages 20-80 years
* spasticity of paretic arm ≤ grade 2 in the Modified Ashworth Scale
* no active medical problems such as fever, pneumonia, or scabies

Exclusion Criteria:

* brainstem or cerebellar stroke
* epilepsy history, including photosensitive epilepsy
* previous or active heart diseases, such as myocardial infarction or angina
* visuospatial problems related to stroke, such as hemianopia or hemineglect
* paretic upper limb reaches Brunnstrom recovery stage VI
* severe aphasia
* severe cognitive impairment
* poor cooperation with assessments

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Stroke Impact Scale (SIS) 3.0 Questionnaire | Baseline (Pre-intervention at 2 days after enrollment)
  Health-Related Quality of Life
Post-Intervention Change of Stroke Impact Scale (SIS) 3.0 Questionnaire | Change from baseline SIS scores at 18 days after enrollment
  Post-intervention Health-Related Quality of Life
3-Month Follow-Up Change of Stroke Impact Scale (SIS) 3.0 Questionnaire | Change from baseline SIS scores at 92 days after enrollment
  3-month follow-up Health-Related Quality of Life
Post-Intervention of Adverse Events or SAE | 16 days
  Proportion of intervention-related adverse events or SAE

SECONDARY OUTCOMES:
Motricity Index (MI) Upper Extremity Test | Baseline (Pre-intervention) at 2 days after enrollment
  Motor impairment and function
Post-Intervention Change of Motricity Index (MI) Upper Extremity Test | Change from baseline MI scores at 18 days after enrollment
  Post-intervention motor impairment and function
3-Month Follow-Up Change of Motricity Index (MI) Upper Extremity Test | Change from baseline MI scores at 92 days after enrollment
  3-month follow-up motor impairment and function
Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Baseline (Pre-intervention) at 2 days after enrollment
  Motor impairment and function
Post-Intervention Change of Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Change from baseline FMA-UE scores at 18 days after enrollment
  Post-intervention motor impairment and function
3-Month Follow-Up Change of Fugl-Meyer Assessment for Upper Extremity (FMA-UE) | Change from baseline FMA-UE scores at 92 days after enrollment
  3-month follow-up motor impairment and function
Self-Care in Functional Independence Measure (FIM) Instrument | Baseline (Pre-intervention) at 2 days after enrollment
  The FIM is an 18-item instrument measuring a person's level of disability in terms of burden of care in six areas including self-care, continence, mobility, transfers, communication, and cognition. Each of the 18 items is graded on a scale of 1-7 based on level of independence in that item (1 = total assistance required, 7 = complete independence). Six items (eating, grooming, bathing, dressing upper body, dressing lower body, and toileting) of self care will be scored and summed in this study.
Post-Intervention Change of Self-Care in Functional Independence Measure (FIM) Instrument | Change from baseline self-care scores at 18 days after enrollment
  The FIM is an 18-item instrument measuring a person's level of disability in terms of burden of care in six areas including self-care, continence, mobility, transfers, communication, and cognition. Each of the 18 items is graded on a scale of 1-7 based on level of independence in that item (1 = total assistance required, 7 = complete independence). Six items (eating, grooming, bathing, dressing upper body, dressing lower body, and toileting) of self care will be scored and summed in this study.
3-Month Follow-Up Change of Self-Care in Functional Independence Measure (FIM) Instrument | Change from baseline self-care scores at 92 days after enrollment
  The FIM is an 18-item instrument measuring a person's level of disability in terms of burden of care in six areas including self-care, continence, mobility, transfers, communication, and cognition. Each of the 18 items is graded on a scale of 1-7 based on level of independence in that item (1 = total assistance required, 7 = complete independence). Six items (eating, grooming, bathing, dressing upper body, dressing lower body, and toileting) of self care will be scored and summed in this study.
Arm Movement Ratio (AMR) Test | Baseline (Pre-intervention) at 1 day after enrollment
  The AMR, the ratio of arm use duration between the more and less affected arm, is detected and calculated by an accelerometer. The participants are asked to wear one accelerometer (ActiGraph wGT3x-BT, ActiGraph, LLC., Pensacola, FL, USA) on each arm for 7 hours.
Post-Intervention Change of Arm Movement Ratio (AMR) Test | Change from baseline AMR scores at 19 days after enrollment
  The AMR, the ratio of arm use duration between the more and less affected arm, is detected and calculated by an accelerometer. The participants are asked to wear one accelerometer (ActiGraph wGT3x-BT, ActiGraph, LLC., Pensacola, FL, USA) on each arm for 7 hours.
3-Month Follow-Up Change of Arm Movement Ratio (AMR) Test | Change from baseline AMR scores at 93 days after enrollment
  The AMR, the ratio of arm use duration between the more and less affected arm, is detected and calculated by an accelerometer. The participants are asked to wear one accelerometer (ActiGraph wGT3x-BT, ActiGraph, LLC., Pensacola, FL, USA) on each arm for 7 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Min Chen, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chiayi Chang Gung Memorial Hospital, Pozi, Taiwan

IPD SHARING:
Plan to Share IPD: No